CLINICAL TRIAL: NCT04126759
Title: Calibration of a Non-invasive Glucose Measurement Device and Assessment of Its Performance in the Hypoglycemic Range in Patients With Type 1 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RSP Systems A/S (Industry)
Collaborators: Steno Diabetes Center Copenhagen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: RSP-17
Record Dates: First submitted 2019-07-15; First posted 2019-10-15 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Diabetes Mellitus
Keywords: Non-invasive glucose monitoring; Raman spectroscopy
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Protocol 1 (Experimental): The subjects enrolled in this protocol will dedicate 33 days of home-based measurement and two days for in-clinic measurements. For reference measurements, subjects will be equipped with a BG-meter (Contour Next One, Ascenia). Optical measurements are collected with the IMD. Each day of measurements consists of four sessions each comprising two capillary blood glucose measurement with a BG-meter and two IMD measurements. IMD measurements will be performed using the thenar of the right hand of the subject.
  Interventions: Device: P0.3

INTERVENTIONS:
Device: P0.3 — Subjects will perform daily measurements on the IMD (Prototype 0.3) for 35 days.

SUMMARY:
This clinical study has been launched to collect spectral Raman data and reference measurements to establish and validate a calibration model for the device during daily glycemic fluctuations and evaluate analytical performance of device in the hypoglycemic range. The study is a combined home-based and in-clinic study where subjects will attend the clinic two times.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects between 18 and 40 years of age.
* Diagnosed with type 1 diabetes mellitus.
* Uses an insulin pen or pump.
* Hb1Ac > 55 mmol/mol at baseline visit.
* Skin phototype 1-4 according to Fitzpatrick skin tone scale.
* Willing to perform a minimum of 8 finger sticks per day during the study for the home-based study and approximately 16 finger sticks for the in-clinic study days.
* Willing to have a peripheral venous catheter inserted.
* Willing to provide written signed and dated informed consent.

Exclusion Criteria:

* Breastfeeding, pregnant, attempting to conceive or not willing and able to practice birth control according to approved contraceptives from NCA during the study execution (applicable to female subjects only).
* Subjects not able to understand and read Danish.
* Inability to comply with the study procedures as described by the study protocol, according to the opinion of the investigator.
* Subject is not able to hold hand/arm steadily (including tremors and Parkinson's Disease).
* Reduced circulation in hand. "Allen's test" is used for assessing hand circulation to evaluate occurrence of reduced blood.
* Extensive skin changes, tattoos or diseases on probe application site (thenar) that could interfere with the accuracy of the interstitial glucose measurements.
* Known allergy to medical grade alcohol.
* Having active cancer treatment and/or use tetracyclines and other medication / topical agents known to increase photosensitivity in skin.
* Medical history or any condition that may, in the opinion of the Investigator, compromise the subject's ability to participate
* Concomitant medical condition which could present a risk to the safety or welfare of the subject or study staff.
* Diagnosed with cardiovascular diseases.
* Subjects currently enrolled in another study.
* Radiotherapy for the past six months.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Generation of predictive algorithms for determining blood glucose levels | 12 months
  Collected spectral raman data will found the development of predictive algorithms for glucose determination.
Validation of predictive algorithms for determining blood glucose levels | 12 months
  Performance of predictive models will be evaluated using the consensus error grid.Unified Performance (ISUP), Mean Absolute Relative Difference (MARD) and Consensus Error Grid (CEG) distribution.

SECONDARY OUTCOMES:
Risk/benefit analysis | 12 months
  Support of a favorable risk/benefit analysis based on reported Adverse Device Effects and Serious Adverse Device Effects.
Number of encountered Device Deficiencies | 12 months
  Evaluation of Device Deficiencies with respect to identity, quality, durability or reliability, including malfunctions, use errors and inadequate labeling.

CONTACTS AND LOCATIONS:
Overall Officials: Kirsten Nørgaard, Principal Investigator — Steno Diabetes Center Copenhagen
Locations (1):
- Steno Diabetes Center Copenhagen (SDCC), Gentofte Municipality, Denmark

IPD SHARING:
Plan to Share IPD: No